CLINICAL TRIAL: NCT07337148
Title: Increasing Mental Health Literacy and Peer Support Among Caregivers: An Electronic Painting and Peer Supportive (EPPS) Platform
Brief Title: Mental Health Literacy and Peer Support Among Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Professor, Associate Head (Research), The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20230421001
Record Dates: First submitted 2025-08-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mental Health
Keywords: Peer support; Caregivers; Electronic painting; Mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We will recruit 700 caregivers through 30 units of NGOs over 2 years. Caregivers can join a 2-hour face-to-face workshop and learn how to download the EPPS system, all the features of the EPPS system, how to draw electronic paintings, share the paintings, and seek help from others via the system. In the workshop, caregivers are given opportunities to meet the designated caregiver support team member in person before they go for online interaction in the coming 8 weeks. The caregivers will also have hands-on practice (how to draw and share the paintings). This is to ensure the caregivers know how to use the EPPS system before they go home. Trained university students or volunteers from NGOs (about 80-100) will assist caregivers download and use the system in the workshop. If the caregivers are not able to join the workshop, the Project Team will share the Powerpoint (that shows how to download and use the system) with them. Telephone advice will be given to these caregivers to ensure t
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): Caregivers in the IG will use the e-painting and e-chat features in the EPPS system for 8 weeks (at the same time, they will continue to receive the usual supportive service to caregivers in the NGOs).
  Interventions: Behavioral: Electronic Painting and Peer Supportive
- Control group (CG) (Active Comparator): The caregivers in the CG will receive e-chat and usual care (the usual supportive service to caregivers in the NGOs). After 8 weeks, the caregivers in the CG will be given opportunities to use the e-painting in the EPPS system.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Electronic Painting and Peer Supportive — The EPPS system consists of five features: 1) electronic painting (e-painting); 2) picture sharing; 3) e-chat; 4) mood self-assessment and 5) announcement. The IG is given all the five features for 8 weeks. At the same time, they will continue to receive the usual supportive service to caregivers in the NGOs.
  Arms: Intervention Group (IG)
Behavioral: Usual Care — The CG receives usual supportive service to caregivers in the NGOs and get access to e-chat in the EPPS system.
  Arms: Control group (CG)

SUMMARY:
This study aims to assess the efficacy of an electronic painting and peer support platform on help seeking behaviour and emotion (depression, anxiety and stress) among caregivers. This is a 2-arm randomized controlled trial with 700 caregivers being randomized to intervention group (IG) or control group (CG). Participants of the IG will use the EPPS system for 8 weeks, making electronic paintings, sharing the paintings with peers, self-assessing emotion and use the provided list to seek for help if necessary. At the same time, they will continue to receive the usual supportive service to caregivers in the NGOs, while the caregivers in the CG will receive e-chat and usual care (the usual supportive service to caregivers in the NGOs). After 8 weeks, the caregivers in the CG will be given opportunities to draw paintings in the EPPS system. All caregivers are invited to complete an online survey at Week 0 (before they use the system), Week 8 (immediately after the system use) and Week 12 (4 weeks after the system use). 30 to 40 caregivers will be invited to attend focus group interviews to indicate their comments and views on the use of the EPPS system after Week 8. Such qualitative data collection will be ceased when no new comments is received. The findings of the study will provide evidence of technology use in supporting caregivers for help seeking and reducing depression, anxiety and stress.

DETAILED DESCRIPTION:
During the 8-week period, caregivers are encouraged to draw paintings. There is no fixed frequency for making the paintings but they are recommended to draw at least one painting per week. Caregivers could draw the electronic paintings at any time when they are free. They could share the paintings with friends or peers in the group. 10-12 caregivers will be gathered as a small group for interaction (supported by a supportive team member). During this period, the supportive team members will announce a theme for drawing each week. Caregivers can self-assess their mental health status by using the validated scale, Depression, Anxiety and Stress Scale (DASS-8) which is installed in the EPPS system at Week 0, Week 8 and Week 12. At any time, they draw the painting, caregivers can self-assess their mood by completing PHQ-2. Caregivers can look for the available mental health support services (shown in the system) and seek help, if necessary. They would also approach the facilitators if they need help. On the other hand, the supportive team members will also monitor the mental health assessment scores and make referral to the professionals if necessary.

Study design. A randomized controlled trial with focus group interviews with caregivers and members of supportive team will be used to assess the efficacy of the EPPS system. Caregivers will be randomly assigned to intervention group (IG) and control group (CG). Caregivers in the IG will use the EPPS system for 8 weeks (at the same time, they will continue to receive the usual supportive service to caregivers in the NGOs) while the caregivers in the CG will receive usual care (the usual supportive service to caregivers in the NGOs). After 8 weeks, the caregivers in the CG will be given opportunities to use the EPPS system. All caregivers are invited to complete an online survey at Week 0 (before they use the system), Week 8 (immediately after the system use) and Week 12 (4 weeks after the system use). 30 to 40 caregivers will be invited to attend focus group interviews to indicate their comments and views on the use of the EPPS system after Week 8. Such qualitative data collection will be ceased when no new comments is received (data is saturated).

Outcome measures in the evaluation: Attitudes Toward Seeking Professional Psychological Help-Short Form (ATSPPH-SF) (primary outcome). It consists of 10 items measuring the propensity for seeking help for mental disorders. A 4-point Likert scale ranging from "0=disagree" to "3=agree" is used as the response options. Total score, ranging from 0 to 30, is calculated by summing up all the items - higher scores indicate higher propensity to seek help. There are two subscales (1) openness to seeking treatment and (2) need in seeking treatment in this instrument. Other outcome measures include: DASS-8, WHO-5 [9], Chinese version of Zarit Burden Interview (CZBI-short), Modified Medical Outcome Study Social Support Survey (mMOS-SS) and PHQ-2 [12]. The DASS-8 is the shortest version of the DASS-21. It is composed of three subscales: depression (three items, e.g., felt that I had nothing to look forward), anxiety (three items, e.g., felt close to panic), and stress (two items, e.g., was using a lot of my mental energy) (36, 38). The minimum score of the DASS-8 and its subscales is 0, while the maximum scores are 24, 9, 9, and 6, respectively. Cronbach alpha = 0.933, and its correlation with DASS-21 is 0.977.

The sample size required for evaluating the efficacy of the EPPS system (using RCT) is calculated with reference to ATSPPH-SF (primary outcome). In a previous study, 65 adults changed their help seeking behaviour (total score of ATSPPH-SF) after watching a short video, and the mean ATSPPH-SF score was 18.1 (SD = 4.3) at pre-test and 19.4 (SD = 3.8) at post-test. The effect size of this e-learning was 0.46. Using a conservative approach, we assume the learning from the AIMHS system has small effect size (=0.3). Using G*Power 3.1.9.4, we assume an effect size of 0.3 with 90% power, two-tailed 5% significance, and 1:1 allocation ratio, the estimated sample size required is 382 (191 per group). Assuming 55% attrition, we intend to recruit about 700 caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers who take care of elderly, disabled, demented, or mentally ill persons
* Able to speak Cantonese
* Live in Hong Kong

Exclusion Criteria:

* currently suffer from severe acute illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Attitudes Toward Seeking Professional Psychological Help-Short Form (ATSPPH-SF) | T0 (baseline), T1 (after the intervention at Week 9), and T2 (week 12)
  It consists of 10 items measuring the propensity for seeking help for mental disorders. A 4-point Likert scale ranging from "0=disagree" to "3=agree" is used as the response options. Total score, ranging from 0 to 30, is calculated by summing up all the items - higher scores indicate higher propensity to seek help. There are two subscales (1) openness to seeking treatment and (2) need in seeking treatment in this instrument.

SECONDARY OUTCOMES:
DASS-8 | T0 (baseline), T1 (after the intervention at Week 9), and T2 (week 12)
  The DASS-8 is the shortest version of the DASS-21. It is composed of three subscales: depression (three items, e.g., felt that I had nothing to look forward), anxiety (three items, e.g., felt close to panic), and stress (two items, e.g., was using a lot of my mental energy) (36, 38). The minimum score of the DASS-8 and its subscales is 0, while the maximum scores are 24, 9, 9, and 6, respectively. Cronbach alpha = 0.933, and its correlation with DASS-21 is 0.977
WHO-5 | T0 (baseline), T1 (after the intervention at Week 9), and T2 (week 12)
  The WHO-5 is a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.
Chinese version of Zarit Burden Interview (CZBI-short) | T0 (baseline), T1 (after the intervention at Week 9), and T2 (week 12)
  The Chinese version of the Zarit Burden Interview (CZBI) is a tool used to assess the burden experienced by caregivers of individuals with dementia. It has a full 22-item version and a shorter 12-item version, known as the CZBI-Short, which is specifically validated for use with Cantonese-speaking caregivers in clinical and social care settings.
Modified Medical Outcome Study Social Support Survey (mMOS-SS) | T0 (baseline), T1 (after the intervention at Week 9), and T2 (week 12)
  The Modified Medical Outcomes Study Social Support Survey (mMOS-SS) is a shortened, 8-item version of the original 19-item Medical Outcomes Study Social Support Survey (MOS-SS). It assesses an individual's perception of social support, specifically focusing on emotional and instrumental (tangible) support. The abbreviated version is designed to be more time-efficient while maintaining the core structure of the original survey and identifying potential deficits in social support.
PHQ-2 | T0 (baseline), T1 (after the intervention at Week 9), and T2 (week 12)
  Patient Health Questionnaire-2, is a brief two-question screening tool used to identify individuals who may be experiencing symptoms of depression. It is a subset of the PHQ-9 and focuses on the frequency of depressed mood and anhedonia (loss of interest or pleasure) over the past two weeks.
Multidimensional Scale of Perceived Social Support (MSPSS) | T0 (baseline), T1 (after the intervention at Week 9), and T2 (Week 12)
  The MSPSS has 12 items measuring perceived social support from 3 sources: family, friends and a significant other. Items were rated on a 7-point Likert scale. The MSPSS total score ranges 7 - 84 and scores of the three dimensions range 4 -24, with higher scores indicating higher levels of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Leung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liang X, Guo Q, Luo J, Li F, Ding D, Zhao Q, Hong Z. Anxiety and depression symptoms among caregivers of care-recipients with subjective cognitive decline and cognitive impairment. BMC Neurol. 2016 Oct 3;16(1):191. doi: 10.1186/s12883-016-0712-2. PMID 27716098
- [Result] Ma M, Dorstyn D, Ward L, Prentice S. Alzheimers' disease and caregiving: a meta-analytic review comparing the mental health of primary carers to controls. Aging Ment Health. 2018 Nov;22(11):1395-1405. doi: 10.1080/13607863.2017.1370689. Epub 2017 Sep 5. PMID 28871796
- [Result] Xu XY, Leung D, Leung AYM, Kwan RYC, Liang TN, Chai AJ. "Am I entitled to take a break in caregiving?": Perceptions of leisure activities of family caregivers of loved ones with dementia in China. Dementia (London). 2022 Jul;21(5):1682-1698. doi: 10.1177/14713012221093879. Epub 2022 Apr 28. PMID 35481765
- [Result] Leung AYM, Cheung T, Fong TKH, Zhao IY, Kabir ZN. The Use of an Electronic Painting Platform by Family Caregivers of Persons with Dementia: A Feasibility and Acceptability Study. Healthcare (Basel). 2022 May 9;10(5):870. doi: 10.3390/healthcare10050870. PMID 35628007
- [Result] Confectioner K, Currie A, Gabana N, van Gerven N, Kerkhoffs GMMJ, Gouttebarge V. Help-seeking behaviours related to mental health symptoms in professional football. BMJ Open Sport Exerc Med. 2021 May 17;7(2):e001070. doi: 10.1136/bmjsem-2021-001070. eCollection 2021. PMID 34055385
- [Result] Ali AM, Alameri RA, Hendawy AO, Al-Amer R, Shahrour G, Ali EM, Alkhamees AA, Ibrahim N, Hassan BH. Psychometric evaluation of the depression anxiety stress scale 8-items (DASS-8)/DASS-12/DASS-21 among family caregivers of patients with dementia. Front Public Health. 2022 Oct 25;10:1012311. doi: 10.3389/fpubh.2022.1012311. eCollection 2022. PMID 36388286
- [Result] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Result] Tang JY, Ho AH, Luo H, Wong GH, Lau BH, Lum TY, Cheung KS. Validating a Cantonese short version of the Zarit Burden Interview (CZBI-Short) for dementia caregivers. Aging Ment Health. 2016 Sep;20(9):996-1001. doi: 10.1080/13607863.2015.1047323. Epub 2015 May 27. PMID 26016419
- [Result] Moser A, Stuck AE, Silliman RA, Ganz PA, Clough-Gorr KM. The eight-item modified Medical Outcomes Study Social Support Survey: psychometric evaluation showed excellent performance. J Clin Epidemiol. 2012 Oct;65(10):1107-16. doi: 10.1016/j.jclinepi.2012.04.007. Epub 2012 Jul 20. PMID 22818947
- [Result] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691

DOCUMENTS (1):
  • Informed Consent Form (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT07337148/ICF_000.pdf